CLINICAL TRIAL: NCT04184024
Title: A Comparison of the Effectiveness of Massage and Kinesio Taping on Pain, Range of Motion, Disability and Quality of Life in Patients With Chronic Neck Pain
Brief Title: A Comparison of the Effectiveness of Massage and Kinesio Taping in Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/10/03
Record Dates: First submitted 2019-11-30; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Neck Pain
Keywords: neck pain, massage, kinesio tape,
MeSH Terms: conditions — Neck Pain | interventions — Massage; Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Active Comparator): Patients in this group were applied to massage plus neck stabilization exercise.
  Interventions: Other: Massage; Other: Neck stabilization exercise
- Kinesio taping group (Active Comparator): Patients in this group were applied to Kinesio taping plus neck stabilization exercise.
  Interventions: Other: Kinesio tape; Other: Neck stabilization exercise

INTERVENTIONS:
Other: Massage — Soft tissue massage known as "Swedish massage" technique was applied to the neck area for 20 minutes. This massage was carried out 3 days a week for 4 weeks (12 sessions) by the supervisor physiotherapist.
  Arms: Massage group
Other: Kinesio tape — Patients were taped according to the Kenzo Kase's Kinesio Taping Method by an experienced physical therapist. The application was carried out in a relaxed sitting position. Y banding with extensor muscles on the back of the neck with muscle technique, I banding with the upper trapezius with muscle technique and I banding with ligament technique to the middle region of the neck were performed.
  Arms: Kinesio taping group
Other: Neck stabilization exercise — Neck stabilization exercise was performed in stages with gradual progression according to the stages of motor learning and sensory-motor integration, namely, static, dynamic, and functional. The program started with postural training and then the cervical bracing technique with the activation of deep neck flexors for NSE was performed. The patients were asked to maintain a neutral spine during the exercises and throughout the day as much as possible. The difficulty and variety of exercises were increased weekly. It was carried out 3 days a week for 4 weeks (12 sessions) by the supervisor physiotherapist.

SUMMARY:
This study aimed to compare the effectiveness of massage and Kinesio taping on pain, range of motion, disability and quality of life in patients with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a common condition, affecting 30% to 50% of the general population, and is most prevalent in middle age.33 It is usually accompanied by a substantial effect on daily life, resulting in an extensive use of health care resources.

Several physical therapy applications such as massage therapy, kinesio taping, thermal and electrophysiological agents, hydrotherapy/spa therapy, and therapeutic exercises especially neck stabilization exercise are used to manage FM. Both massage therapy and kinesio taping have a favorable effect on clinical symptoms. However, it is not clear which method is more effective. Therefore, this study aimed to compare the effectiveness of massage and Kinesio taping on pain, range of motion, disability and quality of life in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* having generalized neck pain for more than 3 months,
* being volunteer

Exclusion Criteria:

* pregnancy,
* inflammatory rheumatologic diseases,
* malignity,
* structural deformity,
* previous surgery related to the cervical spine,
* cervical spinal stenosis,
* being allergic to Kinesio tape
* severe psychological disorder,
* any intervention that included exercise or physical therapy in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Pain Level (Visual Analog Scale) | change from baseline at 4 weeks
  The pain level was assessed with the Visual Analog Scale, which consists of a horizontal line of 10 cm in length. For pain level assessment, "0" defines "no pain" and "10" defines "unbearable pain''. The participants are asked to mark the intensity of their pain level.

SECONDARY OUTCOMES:
Turkish of the Short Form-36 | change from baseline at 4 weeks
  The quality of life was assessed with the Turkish of the Short Form-36 (SF-36). The SF-36 consists of 36 questions: physical functioning (10 items), role limitations due to physical health (4 items), bodily pain (2 items), social functioning (2 items), vitality (4 items), role limitations due to emotional health (3 items), mental health (5 items), general health perceptions (5 items) and changes in health over time (1 item, not included in the final score). The SF-36 score ranges from 0 (the worst score) to 100 (the best score). Thus, higher scores indicate better health. The participants are asked to fulfill the questionnaire.
Turkish version of Neck Disability Index | change from baseline at 4 weeks
  The disability level was measured with the Turkish version of Neck Disability Index (NDI). It consists of 10 sections which include the severity of pain, personal care, lifting, reading, headache, concentration, work-life, driving, sleeping and leisure activities. There are 6 responses for each section, scored 0 (no pain and no functional limitation) and 5 (worst pain and maximum limitation). The total score ranges from 0 to 50. Patients were asked to select the most appropriate option for each section.
Range of Motion | change from baseline at 4 weeks
  The range of motion of the neck joints of the patients was measured with a clinical goniometer (Baseline Evaluation Tools, USA) for flexion, extension, lateral flexion and rotation movements while sitting upright on the stool.

CONTACTS AND LOCATIONS:
Overall Officials: seyda toprak celenay, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No